CLINICAL TRIAL: NCT06141928
Title: Comparison of Three Different Surgical Approaches on the Functional Outcome After Total Hip Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinic for Orthopedics Lovran (Other)
Collaborators: Special Hospital for Orthopedics Biograd na Moru (Unknown)
Responsible Party: Principal Investigator, Antea Buterin, Head of Department, Clinic for Orthopedics Lovran
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Clinic OL
Record Dates: First submitted 2023-02-20; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Total Hip Arthroplasty; Functional Recovery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional Recovery (Other)
  Interventions: Other: Functional recovery analysis

INTERVENTIONS:
Other: Functional recovery analysis — Functional recovery analysis with force evaluator & tester

SUMMARY:
This study aimed to determine differences in functional recovery after total hip arthroplasty between a group of patients operated on using a direct lateral approach, an anterolateral minimally invasive approach, and a posterior approach to the hip joint.

Arthroplasty is the most commonly performed surgical procedure in orthopedics and is also considered the gold standard for treating the final stage of osteoarthritis. There are several different approaches, but there are still conflicting studies that talk about the benefits of a particular approach. There is an insufficient number of scientific, prospective studies that monitor the basic functional and rehabilitation parameters, which are also indicators of the success of the performed procedure.

ELIGIBILITY:
Inclusion Criteria:

* hip osteoarthritis

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional recovery after total hip arthroplasty / Range of motion | 2 years
  Investigators analyze active and passive range of motion (ROM) measured in degrees.
Functional recovery after total hip arthroplasty / Walking speed | 2 years
  Investigators analyze walking speed in seconds for the 50 meters long walk.
Functional recovery after total hip arthroplasty / Harris Hip Score | 2 years
  Investigators take a questionnaire (Harris Hip Score, HHS), the maximum point is 100.
Functional recovery after total hip arthroplasty / Hip abductors strength | 2 years
  Investigators analyze hip abductors strength measured with a dynamometer in kilograms (kg).

CONTACTS AND LOCATIONS:
Overall Officials: Antea Buterin, MD, Principal Investigator — Clinic OL
Locations (1):
- Clinic for Orthopeadics and Traumatology Lovran, Lovran, Primorje-Gorski Kotar County, Croatia

IPD SHARING:
Plan to Share IPD: Undecided